CLINICAL TRIAL: NCT05492188
Title: Targeted Spinal Cord Plasticity for Alleviating SCI-related Neuropathic Pain
Brief Title: Neuropathic Pain and Operant Conditioning of Cutaneous Reflexes After SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aiko Thompson, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118771; CDMRP-SC210118 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain; Neurological Injury; Pain
Keywords: Neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Trauma, Nervous System; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Operant Conditioning of Cutaneous Reflexes (Experimental): Each participant completes 6 baseline sessions and 30 conditioning sessions. In each of the 30 conditioning sessions, while the participant is standing nerves in the lower leg and ankle are stimulated to activate the reflex. The participant attempts to change the reflex activity based on visual feedback. In this way the cutaneous reflex (skin reflex) will be changed to decrease neuropathic pain resulting from spinal cord injury.
  Interventions: Behavioral: Operant Conditioning of Cutaneous Reflexes

INTERVENTIONS:
Behavioral: Operant Conditioning of Cutaneous Reflexes — This is a training intervention in which people with a spinal cord injury are trained to change (increase or decrease) the activity of a certain spinal reflex. By changing this reflex, it is hypothesized that individuals can reduce pain due to spinal cord injury.

SUMMARY:
The purpose of the second part of the study is to examine the effect of reflex training in the leg to decrease neuropathic pain. For this, the researchers are recruiting 15 individuals with neuropathic pain due to spinal cord injury to participate in the reflex training procedure. The study involves approximately 50 visits with a total study duration of about 6.5 months (3 months for baseline and training phases followed by 1 month and 3 month follow-up visits).

DETAILED DESCRIPTION:
As part of the larger study of the relationship between reflexes in the leg and the presence of neuropathic pain, the researchers are also recruiting 30 individuals with spinal cord injury (SCI) total, 15 individuals with neuropathic pain due to SCI and 15 individuals without neuropathic pain. For this portion of the study, there are 2 visits. The first visit will examine cutaneous reflexes in the leg. During the second visit, the study team will assess sensation in the leg and administer questionnaires about pain, functioning, and quality of life. This portion of the study does not involve an intervention.

The study will then recruit 15 individuals who will participate in reflex training, as described in the brief summary.

ELIGIBILITY:
Inclusion Criteria:

1. neurologically stable (>1 year post SCI)
2. medical clearance to participate
3. ability to stand with or without an assistive device for at least 3 minutes at a time
4. expectation that current medication will be maintained without change for at least 3 months (stable use of anti-spasticity medication is accepted)
5. For participants with neuropathic pain, the area of neuropathic pain must include lower leg.

Exclusion Criteria:

1. motoneuron injury
2. known cardiac condition
3. medically unstable condition (incl. pregnancy)
4. cognitive impairment
5. uncontrolled peripheral neuropathy
6. frequent use of electrical spinal stimulation (either transcutaneous or epidural) for pain treatment
7. daily use of electrical stimulation to the leg
8. complete lack of cutaneous sensation around foot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in minimum stimulation intensity required to barely detect the sensation (perceived threshold, perT) | change from baseline to immediately after completing the training protocol, at 1 month follow up and at 3 months follow up
  This is measured by slowly increasing the nerve stimulation and recording the minimum intensity of stimulation at which the participant is barely able to perceive the sensation. A decrease in this threshold would demonstrate improved sensation.
Change in minimum intensity at which the sensation covers the maximum area of skin (radiating threshold, RT) | change from baseline to immediately after completing the training protocol, at 1 month follow up and at 3 months follow up
  This is measured by slowly increasing the nerve stimulation and recording the minimum intensity of stimulation at which the sensation covers the maximum skin area). A decrease in this threshold indicates improved sensation.
Change in minimum intensity at which the stimulus become painful (pain threshold, PainT) | change from baseline to immediately after completing the training protocol, at 1 month follow up and at 3 months follow up
  This is measured by slowly increasing the nerve stimulation and recording the intensity of stimulation at which the stimulation first becomes painful. An increase in this threshold indicates an increased tolerance to pain.
Change in pain as measured by the McGill Pain Questionnaire (MPQ) | Completed at baseline, start of conditioning visits 13, 19, and 25, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  The MPQ is a self-report questionnaire that assesses quality and intensity of pain. Scores range from 0 (no pain) to 78 (severe pain).
Change in neuropathic pain as measured by the Neuropathic Pain Symptom Inventory (NPSI) | Completed at baseline, start of conditioning visits 13, 19, and 25, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  The NPSI is a self-report questionnaire that characterizes neuropathic pain symptom severity. Participants rate different symptoms of neuropathic pain on a scale of 0 (no pain) to 10 (intense pain).

SECONDARY OUTCOMES:
Change in ability to perceive various types of sensations as indicated by Quantitative Sensory Testing (QST) | Completed at baseline, start of conditioning visits 13, 19, and 25, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  The QST is a battery of assessments that measure sensory thresholds for pain, touch, vibration, and hot and cold temperature sensations.
Change in basic functional independence as measured by the Spinal Cord Independence Measure (SCIM III) | Completed at baseline, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  An increase in the the score on the SCIM III indicates increased basic functional independence. This is a self report questionnaire with 19 items in three sub-scales: (1) self-care (6 items, subscore 0-20); (2) respiration and sphincter management (4 items, subscore 0-40); and (3) mobility (9 items, subscore 0-40). The total score ranges from 0-100, with higher scores indicated increase independence.
Change in functional independence as measured by the Functional Independence Measure (FIM) | Completed at baseline, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  An increase in the score on the FIM indicates and increase in functional independence. This 18-item, clinician-reported scale assesses function in 6 areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence).
Change in quality of life as measured by Spinal Cord Injury Quality of Life and Participation Questionnaire (SCI-QOL) | Completed at baseline, after completing 30 conditioning sessions, 1 month follow up, and 3 months follow up
  An increase in score on the SCI-QOL indicates an increase in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Aiko Thompson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT05492188/ICF_000.pdf